CLINICAL TRIAL: NCT07272876
Title: Investigation of the Relationship Between Kinesiophobia, Pain Intensity, and Physical Performance in Elderly Individuals With Musculoskeletal Pain
Brief Title: Kinesiophobia and Physical Function in Elderly With Musculoskeletal Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Zeynep Kaçar Akkoç, Principal Investigator, Istinye University
Other Study IDs: 24-313
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Pain; Physical Performance; Geriatrics; Kinesiophobia
Keywords: musculoskeletal pain; Physical Performance; Geriatrics; Kinesiophobia
MeSH Terms: conditions — Musculoskeletal Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Individuals With Musculoskeletal Pain: This cohort consists of community-dwelling adults aged 65 years and older who are experiencing musculoskeletal pain. Participants in this group present with age-related degenerative musculoskeletal conditions that may affect movement, balance, and functional ability. All individuals in this cohort undergo standardized assessments of kinesiophobia, pain intensity, and physical performance. The cohort reflects a population with chronic musculoskeletal symptoms but without distinctions based on specific diagnoses, treatment exposure, or disease severity.

SUMMARY:
This study aims to investigate how kinesiophobia (fear of movement), pain intensity, and physical performance are related in older adults experiencing musculoskeletal pain. Musculoskeletal pain is highly common in the elderly due to age-related degenerative changes, such as osteoarthritis, chronic low back pain, osteoporosis, and muscle weakness. These conditions often lead to reduced mobility, impaired balance, and limitations in daily living activities. As a result, many older adults may avoid physical activity due to fear of pain or reinjury, which may further decrease their functional capacity.

The primary purpose of this study is to understand whether kinesiophobia contributes to lower physical performance in elderly individuals who have musculoskeletal pain. The study will also examine how pain intensity relates to balance, upper and lower limb strength, and overall functional ability.

Participants aged 65 years and older will complete a set of standard assessments in a single 30-minute session. Kinesiophobia will be measured using the Tampa Scale of Kinesiophobia, a 17-item questionnaire designed to assess fear of movement and avoidance behaviors. Balance will be evaluated with the Berg Balance Scale, which includes 14 tasks commonly performed in daily life. Lower limb strength will be assessed with the 30-Second Sit-to-Stand Test, while upper limb strength will be measured with a handgrip dynamometer.

Understanding these relationships may help clinicians design better rehabilitation programs that reduce fear, improve physical performance, and support healthy aging. The findings of this study may also contribute to strategies for preventing disability and promoting independence in older adults with musculoskeletal pain.

DETAILED DESCRIPTION:
This study is a cross-sectional observational investigation designed to characterize the multidimensional relationship between kinesiophobia, pain intensity, and physical performance in older adults presenting with musculoskeletal pain. Age-related degeneration affecting musculoskeletal tissues-such as reduced muscle cross-sectional area, impaired proprioceptive feedback, decreased bone mineral density, and deterioration in connective tissue elasticity-frequently results in chronic pain syndromes and diminished functional capacity. These physiological changes, combined with psychological factors such as fear of movement, contribute to a cycle of physical inactivity, deconditioning, balance impairments, and functional decline in the geriatric population.

Study Design and Rationale

Kinesiophobia has been identified as a significant psychological construct influencing mobility, pain perception, and functional outcomes in individuals with chronic musculoskeletal conditions. However, evidence regarding its interaction with objective performance-based metrics in geriatric populations remains limited. This study aims to fill this gap by concurrently evaluating kinesiophobia and physical performance using validated assessment instruments within a standardized protocol. The cross-sectional framework allows for analyzing inter-variable associations without the confounding influence of longitudinal adaptations.

Assessment Protocol

All assessments will be conducted in a controlled clinical environment by licensed physiotherapists who have received prior training and standardization instruction for each measurement tool. The evaluation sequence will be fixed for all participants to minimize order effects. Prior to each data collection day, calibration procedures will be performed for the hand dynamometer (e.g., tension verification using manufacturer-approved calibration weights) to ensure measurement reliability.

The assessment battery includes:

Kinesiophobia Evaluation:

The Tampa Scale of Kinesiophobia (TSK), a 17-item self-administered instrument, will be used to quantify fear-avoidance beliefs related to movement and reinjury. Although primarily psychological, TSK scores have been associated with functional mobility and pain chronicity in prior studies.

Balance Assessment:

Functional balance will be measured using the Berg Balance Scale (BBS), consisting of 14 graded tasks that assess static and dynamic postural control. The scale provides a comprehensive assessment of sensorimotor integration, anticipatory and reactive postural adjustments, and functional stability.

Lower Limb Strength and Endurance:

The 30-Second Sit-to-Stand Test (30s-STS) will operationalize lower extremity strength, endurance, and neuromuscular coordination. This test has demonstrated strong reliability in geriatric cohorts and is sensitive to age-related declines in lower limb function.

Upper Limb Strength:

Handgrip strength will be assessed using a Jamar hydraulic dynamometer, which is considered the gold standard for grip strength evaluation due to its high test-retest reliability and minimal operator bias. Measurements will follow the standardized American Society of Hand Therapists (ASHT) protocol.

Data Governance, Quality Control, and Management

Data will be recorded initially onto paper case report forms (CRFs) during assessments and subsequently transcribed into a secure password-protected digital database. The study will incorporate multiple layers of quality assurance:

Range and Consistency Checks: Automatic validation rules will flag values outside expected physiological ranges or inconsistent with related variables (e.g., BBS item scores outside permissible thresholds).

Source Data Verification (SDV): A qualified researcher will perform periodic verification by comparing electronic entries with original CRFs to ensure transcription accuracy.

Audit Trail: All data modifications will be logged, capturing timestamps and user identification.

Data Handling for Missingness: Missing data will be categorized by mechanism (missing completely at random, missing at random, or missing not at random). Based on this classification, either multiple imputation, expectation-maximization techniques, or listwise deletion will be applied.

Sample Size and Statistical Analysis Plan

The study aims to recruit a sample sufficient to detect at least moderate effect sizes (r ≥ 0.30) with 80% power at a significance level of α = 0.05. Sample size estimation is based on correlation analysis using two-tailed testing parameters.

The primary statistical analyses will include:

Descriptive Statistics: Mean, standard deviation, median, and quartiles for continuous variables; frequencies and proportions for categorical descriptors.

Normality Testing: Shapiro-Wilk or Kolmogorov-Smirnov tests to determine distributional characteristics.

Correlation Analyses: Pearson or Spearman correlation coefficients, depending on normality, to explore pairwise associations among kinesiophobia, pain intensity, and physical performance variables.

Multivariable Regression Modeling: Hierarchical linear regression will be conducted to determine the independent contribution of kinesiophobia and pain intensity to each physical performance outcome, controlling for age, sex, and comorbidity burden if necessary.

Assumption Testing: Regression diagnostics will include variance inflation factors (VIFs), residual normality, heteroscedasticity analyses, and influence statistics (e.g., Cook's distance).

Scientific and Clinical Significance

By integrating psychological and biomechanical domains within a single evaluation framework, this investigation aims to elucidate potential mechanistic pathways linking fear-avoidance behavior with objective impairments in physical performance. Identifying these relationships may provide essential insights for designing targeted rehabilitation protocols that address not only physical deficits but also psychological barriers to movement. The findings may also inform clinical decision-making for fall risk reduction, functional independence preservation, and individualized exercise prescription in older adults with musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years of age
* Having musculoskeletal pain
* Having the ability to read, write, and understand Turkish

Exclusion Criteria:

* Presence of any neurological disease
* Presence of a mental health problem that would prevent participation in the study
* Presence of a metabolic disease such as diabetes or hypothyroidism
* Presence of a malignancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants will be community-dwelling older adults recruited from local geriatric outpatient clinics, physiotherapy centers, and community health facilities. The study population will primarily consist of individuals aged 65 years and above who seek evaluation or follow-up care related to musculoskeletal health, mobility, or general functional status within these clinical and community settings.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia Level (Tampa Scale of Kinesiophobia Score) | At a single assessment session (approximately 30 minutes after enrollment).
  Kinesiophobia will be assessed using the Tampa Scale of Kinesiophobia (TSK), a 17-item self-report questionnaire. Each item is scored from 1 (strongly disagree) to 4 (strongly agree), yielding a total score range of 17 to 68.
  Higher scores indicate greater fear of movement and higher levels of avoidance behavior.

SECONDARY OUTCOMES:
Balance Performance (Berg Balance Scale Score) | At a single assessment session (approximately 30 minutes after enrollment).
  Balance will be assessed using the Berg Balance Scale (BBS), which consists of 14 tasks scored from 0 to 4. The total score ranges from 0 to 56, with higher scores indicating better balance and lower fall risk.
Lower Limb Strength and Functional Performance (30-Second Sit-to-Stand Test Repetitions) | At a single assessment session (approximately 30 minutes after enrollment).
  Lower limb strength and functional mobility will be evaluated using the 30-Second Sit-to-Stand Test. The outcome is the total number of full sit-to-stand repetitions completed within 30 seconds.
  Higher repetition counts indicate better lower extremity strength and functional performance.
Upper Limb Strength (Handgrip Dynamometry) | At a single assessment session (approximately 30 minutes after enrollment).
  Upper limb strength will be assessed using a Jamar hand dynamometer. The outcome measure is the maximum grip force (in kilograms) recorded across three trials.
  Higher values indicate greater upper extremity strength.
Pain Intensity (Numeric Rating Scale) | At a single assessment session (approximately 30 minutes after enrollment).
  Pain intensity will be recorded using the Numeric Rating Scale (NRS), in which participants rate their pain from 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate greater pain severity

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kaçar Akkoç, Principal Investigator — Istinye University; Zeynep Kaçar Akkoç, Principal Investigator — zeynep.kacar@stu.istinye.edu.tr
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided